CLINICAL TRIAL: NCT03802279
Title: Study of the Correlation Between the Effort Test, With the Assessment of Peripheral Oxygen Consumption and Cardiac Output in Patients With Acute Rhabdomyolysis Related to a Hereditary Disease of Metabolism, and the Biochemical Flux on Myoblasts: Evaluate the Effort Test as a Therapeutic Monitoring Tool in Acute Rhabdomyolyses
Brief Title: Evaluate the Effort Test as a Therapeutic Monitoring Tool in Acute Rhabdomyolyses
Acronym: EFFORHAB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 180 009; 2018-A01771-54 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-12-06; First posted 2019-01-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Rhabdomyolysis Linked to a Hereditary Disease of Metabolism
Keywords: Rhabdomyolysis linked to a hereditary disease of metabolism; Correlation between the effort test and the severity of the disease and biochemical flux on myoblasts

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Rhabdomyolysis with myoblasts back up: Patients with a rhabdomyolysis linked to a hereditary disease of metabolism who have benefited from a diagnostically muscle biopsy and whose myoblasts are available.
  Patients benefit from an effort test as part of their care.
  Interventions: Other: Effort test; Other: Functional tests on fibroblasts
- Rhabdomyolysis: Patients with a rhabdomyolysis linked to a hereditary disease of metabolism who have benefited or not from a diagnostically muscle biopsy but whose myoblasts are not available.
  Patients benefit from an effort test as part of their care.
  Interventions: Other: Effort test
- Witness patients : effort test: 10 patient-matched healthy controls for age and sex having performed an effort test and cardiac exploration as part of their care.
  Interventions: Other: Effort test
- Witness patients : myoblasts: 6 healthy controls matched by age and sex having performed a muscle biopsy as part of their care and whose myoblasts are kept.
  Interventions: Other: Functional tests on fibroblasts

INTERVENTIONS:
Other: Effort test — Cardiac function:
  Echocardiography: left ventricular ejection fraction and global longitudinal strain will be measured.
  Cardiopulmonary exercise test (CPET): left ventricular stroke volume was assessed noninvasively using a thoracic bioelectrical impedance device : maximal stroke volume at the peak of effort will be considered.
  Peripheral muscle function:
  * CPET: Oxygen uptake (VO2) (and carbon dioxide) output are measured. The slope of the relationship (dQ/dVO2) will be calculated between cardiac output (Q) and VO2 using measurements of Q (using measure of the stroke volume by thoracic bioelectrical impedance device) and VO2 at rest as well as during submaximal and maximal exercise
  * Muscle oxygenation is measured using a near-infrared spectroscopy device.
  * VO2 et Q will be measured : dQ/dVO2 is high in case of oxydation defect; If Q is low because of a concommittant cardiac impairement, the DAV = VO2/Q, and DO = (Q x DAV) / (200 - DAV) will be calculated.
  Groups: Rhabdomyolysis; Rhabdomyolysis with myoblasts back up; Witness patients : effort test
Other: Functional tests on fibroblasts — Functional tests performed on fibroblasts in primary culture, using as tracers of stable isotope-labeled substrates. The metabolites of interest are assayed in mass spectrometry.
  Groups: Rhabdomyolysis with myoblasts back up; Witness patients : myoblasts

SUMMARY:
The prognosis of rhabdomyolyses related to hereditary diseases of metabolism is poor and treatments are only symptomatic. Rhabdomyolysis outbreaks are frequently precipitated by fever and fasting. They are unpredictable. In spite of the care of patient in an intensive care unit, the occurrence of renal failure and heart rhythm disorders explains a significant acute-phase mortality rate. There is an urgent need to understand the pathophysiological mechanisms of rhabdomyolyses related to hereditary diseases of metabolism, in order to identify specific treatments.

Patients with rhabdomyolyses have few clinical signs outside of access. So there is a methodological difficulty in following a treatment test. There is an urgency to identify follow-up parameters in anticipation of new therapies.

The objective of this study is to validate the hypothesis that effort test and cardiac function parameters are usable in the treatment monitoring for patients with acute rhabdomyolysis linked to a hereditary disease of metabolism and thus propose the effort test as an assessment tool for future clinical trials. In order to do so, the correlation between the results of the effort tests, performed to each patient with rhabdomyolysis related to a hereditary disease of metabolism, with the severity of the disease will be evaluated. This study is original because it opens up innovative prospects for monitoring in the field of hereditary diseases of metabolism, with the identification of new monitoring tools.

DETAILED DESCRIPTION:
Rhabdomyolysis is a poorly known symptom associated with the destruction of skeletal muscle cells. The diagnosis of rhabdomyolyses is carried when the dosage of muscle enzymes, in particular creatine phosphate kinase (KPC), is greater than 1000 U/L (normal < 160 U/L).

Rhabdomyolyses may be of viral origin, but fever and viruses are also triggers of genetic diseases. Also, the incidence of genetic rhabdomyolyses, representing 10 to 15% of all rhabdomyolyses, is underestimated. Genetic causes are heterogeneous. They are mainly attributed to hereditary diseases of metabolism, in particular fatty acid oxidation defects, Lipin-1 deficiency, muscle glycogenoses, TANGO2 deficiency, mitochondrial cytopathies and calcium channels anomalies of in particular RYR1.

Whatever the cause, traumatic, infectious or genetic, the rhabdomyolyses cause an alteration of the metabolism of adenosine triphosphate and a deregulation of the ionic channels, with the consequences of an intracytoplasmic calcium release and the destruction of muscle cells.

The prognosis of rhabdomyolyses related to hereditary diseases of metabolism is poor and treatments are only symptomatic. Rhabdomyolysis outbreaks are frequently precipitated by fever and fasting. They are unpredictable. In spite of the care of patient in an intensive care unit, the occurrence of renal failure and heart rhythm disorders explains a significant acute-phase mortality rate. There is an urgent need to understand the pathophysiological mechanisms of rhabdomyolyses related to hereditary diseases of metabolism, in order to identify specific treatments.

The pathophysiological mechanism of rhabdomyolyses related to Lipin-1 deficiency has been identified. Two patients with Lipin-1 deficiency treated in vivo by Hydroxychloroquine (Plaquenil ®, 6 mg/kg/day by one oral intake) rapidly standardized their serum inflammatory profile and corrected their clinical phenotype: Plasma creatine phosphokinase levels, Amount of mitochondrial DNA in plasma, number of myolyses, muscular pain, quality of life. One of these two patients, suffering from cardiac dysfunction already reported in Lipin-1 deficiency (left ventricular ejection fraction or LVEF 45%), significantly and durably improved cardiac function after one month of treatment (LVEF 62%). In addition, his fatigability and sleep disturbances have dramatically improved.

Disruption of mitophagy and immunity could be a common denominator for rhabdomyolyses linked to hereditary diseases of metabolism, which could, despite their heterogeneity, benefit from a common therapeutic approach, Now non-existent. There could be a role of inflammation in rhabdomyolyses outbreaks of metabolic origin and new therapeutic approaches could be imagined as in the Lipin-1 deficiency.

Patients with rhabdomyolyses have few clinical signs outside of access. So there is a methodological difficulty in following a treatment test. There is an urgency to identify follow-up parameters in anticipation of new therapies.

In the Lipin deficiency, an anomaly of the effort tests with measurement of oxygen consumption and cardiac output was characterized. These effort tests were carried out in the context of care, in order to recognize for a given patient whether the practice of sport is a factor triggering rhabdomyolysis.

The objective of this study is to validate the hypothesis that effort test and cardiac function parameters are usable in the treatment monitoring for patients with acute rhabdomyolysis linked to a hereditary disease of metabolism and thus propose the effort test as an assessment tool for future clinical trials. To date, no tests are available for clinical trials. In order to do so, the correlation between the results of the effort tests, performed to each patient with rhabdomyolysis related to a hereditary disease of metabolism, with the severity of the disease will be assessed, including:

1) Metabolic flux on myoblasts, 2) clinical severity (onset of disease, number of rhabdomyolyses, cardiomyopathy), 3) genotype.

This study is original because it opens up innovative prospects for monitoring in the field of hereditary diseases of metabolism, with the identification of new monitoring tools.

ELIGIBILITY:
subjects with metabolic rhabdomyolysis related to a hereditary metabolic disease :

Inclusion Criteria:

* pathology characterized on the biochemical and molecular level
* patients who can make an effort test
* patients who benefited from a diagnostically targeted muscle biopsy with backup of myoblasts (group 1)
* patients who have benefited from a diagnostically targeted muscle biopsy but whose myoblasts are not available (group 2) Exclusion Criteria
* inability or refusal of compliance to the requirements of the research
* patients with contraindications for the effort test in particular heart failure and acute rhabdomyolysis
* Patients without biochemical and/or molecular diagnosis

Criteria for inclusion of witness patients :

* holders of parental authority and/or patients not opposed to the use of their cardio-respiratory analysis results for this study or to the use of their myoblasts for this study
* normal cardio-respiratory analysis results
* normal myoblasts (group 4).

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population to be studied consists of 40 patients with metabolic rhabdomyolyses followed by the centre of reference for metabolic diseases of the child and adult of the Necker Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of cardiac output (Q) | Day 0
  Effort test
Measurement of oxygen consumption (VO2) | Day 0
  Effort test
Calculation of the slope of the relationship heart rate-oxygen consumed (dQ/dVO2) | Day 0
  Effort test
Calculation of the maximum arteriovenous difference (DAV) : DAV=VO2/Q | Day 0
  Effort test
Calculation of maximum muscle diffusion (DM) using the equation of Fick: DM = (Q x DAV)/(200-DAV) | Day 0
  Effort test
Peripheral muscular oxygenation | Day 0
  Measurement of peripheral muscular oxygenation during the effort test.
Systolic ejection volume at the peak of the effort during the effort test | Day 0
  Evaluation of cardiac performance by the value of the systolic ejection volume at the peak of the effort.
  The systolic ejection volume is measured beat per beat during the effort test.
Ejection fraction of the left ventricle | Day 0
  Measurement of the ejection fraction of the left ventricle in Simpson biplane and the longitudinal strain of the left ventricle in echocardiography.
Metabolic pathways of myoblasts | From study start until 26 months
  Myoblasts will be incubated in the presence of stable isotope-labeled tracers. The natural metabolites labelled with stable isotopes will be dosed. The acylcarnitines will be dosed on a mass spectrometer. The Krebs cycle intermediates will be measured in gas chromatography coupled with mass spectrometry.

SECONDARY OUTCOMES:
Presence of cardiomyopathy | Day 0
  Clinical severity of rhabdomyolysis linked to a hereditary disease of metabolism.
Age of onset of disease (neonatal, < 2 years, 2 - 10 years, > 10 years) | Day 0
  Clinical severity of rhabdomyolysis linked to a hereditary disease of metabolism.
Number of acute episodes of rhabdomyolyses | Day 0
  Clinical severity of rhabdomyolysis linked to a hereditary disease of metabolism.
Character of mutations nonsense or missense of the hereditary disease of metabolism | Day 0
  Genotypic severity of rhabdomyolysis linked to a hereditary disease of metabolism.
  Information available in the patient medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Pascale de Lonlay, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Antoine Legendre, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Florence Habarou, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Caroline Tuchmann-Durand, Pharm. D, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

REFERENCES:
- [Background] Imbard A, de Calbiac H, Le Guillou E, Laforet P, Schiff M, Brassier A, Thevenet E, Pontoizeau C, Lefrere B, Ottolenghi C, Lebigot E, Gaignard P, Gobin S, Acquaviva-Bourdain C, Benoist JF, Tuchmann-Durand C, Legendre A, de Lonlay P. Circulatory response to exercise relative to oxygen uptake assessed in the follow-up of patients with fatty acid beta-oxidation disorders. J Inherit Metab Dis. 2025 Jan;48(1):e12819. doi: 10.1002/jimd.12819. Epub 2024 Dec 9. PMID 39648745